CLINICAL TRIAL: NCT02122640
Title: Evaluation of Acute Cardiogenic Dyspnoea With Thorax Echography and Pro-BNP in the Emergency Department
Acronym: ECO/TOR
Status: Completed | Type: Observational
Sponsor: Comitato Etico di Area Vasta Sud Est (Other)
Responsible Party: Principal Investigator, Marcellopastorelli, Pastorelli, Comitato Etico di Area Vasta Sud Est
Other Study IDs: ECO/TOR
Record Dates: First submitted 2014-04-23; First posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Acute Heart Failure

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
LUNG ULTRASOUND IN THE MANAGEMENT OF DISPNEIC PATIENTS IN EMERGENCY DEPARTMENT

Introduction

This is a prospective randomized trial realized in the Emergency Department of the University Hospital of Siena, Italy.

Dyspnea is one of the most common causes worldwide of admission to the Emergency Department (ED) and acute heart failure (AHF) is a major cause of serious morbidity and death in such population, above all in elderly patients. Incidence rate is signiﬁcantly higher in men than in women, in Europe it increases with age from 1.4/1000 person-years in subjects aged 55-59 years to 47.4/1000 person-years in those aged 90 years or older. The age-adjusted prevalence of AHF in the United States averages 36 cases per 100,000 of the population and accounts for 10,000 deaths annually.

In clinical practice this symptomatology is usually investigated in the pre-hospital phase only with history and physical examination; in the ED blood gas analysis (BGA), laboratory tests and chest X-rays can be performed as primary exams. BNP and NT pro-BNP are now considered reliable biochemical markers to distinguish cardiogenic from pulmonary etiology, both for their diagnostic and prognostic value. On the other hand, these biomarkers are affected by a "grey zone" of uncertainty, they are not available in all hospitals and their dosage samples are expensive: thus we propose other tools to support the diagnostic process.

DETAILED DESCRIPTION:
THE RATIONALE OF THE STUDY

It is widely reported in literature that ultrasound can identify the presence of interstitial and pulmonary alveolar syndrome by comet tail artifact with good sensitivity and specificity. This is an easy technique to perform and interpret, readily available and repeatable over time and executable bedside even in emergency situations. The execution of this investigative technique in the ED and also in a pre-hospital setting would provide additional and reliable information for patients with dyspnea, so favoring rapid identification of the etiology.

Accepting these observations, lung ultrasound (LUS) could have a central role in the evaluation of patients with shortness of breath in ED. Even the LUS in many studies has been considered useful for detecting pulmonary alterations, there are few data regarding its utilization in clinical practice and there is a lack of evidences concerning validated operative protocols. On this basis, it was decided to evaluate the employment of LUS in the ED with a structured and practical protocol.

ETHICAL ASPECTS

This study will be conducted according to Helsinki Declaration and i twill be approved by our Local Ethics Committee.

AIMS OF THE STUDY

The main aim of this study was to analyze if lung ultrasound (LUS) could be a useful tool for the early identification of heart failure in patients presenting to ED for dyspnea.

The secondary objective was to identify a protocol model for the management of acute dyspnea on the basis of lung ultrasound pattern when added to other validated diagnostic tools.

INCLUSIONS CRITERIA

All the patients admitted to our Emergency Department from January 2011 to February 2013 with acute non-traumatic dyspnea. We included patients carried by ambulance and patients who came autonomously.

EXCLUSIONS CRITERIA

Age <18 years

Post-traumatic dyspnea

METHODS

After triage, standardized diagnostic work-up included: 1) brief patient history (age, gender, symptoms, medical history); 2) Vital Parameters (Blood Pressure, Heart Rate, Arterial Oxygen Saturation, Respiratory Rate, Body Temperature); 3) 12 lead EKG; 4) Standard laboratory assessment (NT-proBNP - ECLIA, Roche Methodics®, Creatinine, BUN, C-Reactive Protein, Full Blood Count, Electrolytes); 5) Blood Gas Analysis. Data were collected and stored in a database.

An independent operator performed LUS right after the admission (unaware of patient history and vitals), then the attending physician acquired full medical history, Physical Examination (according to Boston Criteria for Heart Failure) and requested Chest X-Ray. Echocardiography was performed in order to validate heart failure diagnosis even if it was not considered in our protocol because not available 24h/day in our Emergency Department. All LUS operators were emergency physicians trained in LUS.

Lung Ultrasound We used Esaote MyLab30™ and MyLab70™ Ultrasound with Variable-Band Convex Array (3,5-5 MHz). Six transversal scans for each hemithorax (second and fourth intercostal space on the hemiclavear line, anterior axillar line, middle axillar line, see Figure 1). Basal scans of the lung were sampled in order to identify pleural effusions.

We chose this anterior approach for the difficulties related to a complete evaluation of the chest in case of severe dyspnea and non-collaborative patients.

B-lines are defined as vertical, hyperechogenic, reverberation artifacts that arise from the pleural line to the bottom of the screen and moving synchronously with lung sliding; a positive region is defined by the presence of three or more B-lines in a longitudinal plane between two ribs. Acute interstitial pulmonary syndrome was defined, according to the International Consensus Conference on LUS, as the presence of two or more positive regions in each hemithorax.

Diagnostic Outcome (Reference Standard) Since a uniform reference test is lacking for acute heart failure, we chose to use a consensus diagnosis as formal reference standard, in analogy with earlier studies and as recommended by recent diagnostic research guidelines. An independent panel of experts (made up of two cardiologists and one senior emergency physician) judged all the collected data for each patient to determine the final diagnosis.

The panel of experts assessed acute heart failure diagnosis following the criteria and approach outlined by the ESC Heart Failure Guidelines.

LENGHT OF THE STUDY

From January 2011 to February 2013

DATA COLLECTION

Data collection form included:

Personal data Medical hystory VItals signs; ECG; BGA; Medical Examination; Standard Blood Test plus NT pro-BNP; Chest X-ray; Echocardiography; Lung Ultrasound

STATISTICAL ANALYSIS

Edited to Prof. Cevenini.

ELIGIBILITY:
Inclusion Criteria:

All the patients admitted to our Emergency Department from January 2011 to February 2013 with acute non-traumatic dyspnea. We included patients carried by ambulance and patients who came autonomously.

Exclusion Criteria:

* Age <18 years

Post-traumatic dyspnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients admitted to our Emergency Department from January 2011 to February 2013 with acute non-traumatic dyspnea. We included patients carried by ambulance and patients who came autonomously.
Sampling Method: Non-Probability Sample
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic Outcome (Reference Standard) | 1 day
  Since a uniform reference test is lacking for acute heart failure, we chose to use a consensus diagnosis as formal reference standard, in analogy with earlier studies and as recommended by recent diagnostic research guidelines. An independent panel of experts (made up of two cardiologists and one senior emergency physician) judged all the collected data for each patient to determine the final diagnosis.
  The panel of experts assessed acute heart failure diagnosis following the criteria and approach outlined by the ESC Heart Failure Guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Senese, Siena, Siena, Italy